CLINICAL TRIAL: NCT01021410
Title: Serum Acetaminophen-Cysteine (APAP-cys) Adduct Concentrations After 16 Days of Acetaminophen Dosing
Brief Title: Acetaminophen-Protein Adduct Resolution
Acronym: AR
Status: Completed | Type: Observational
Sponsor: Denver Health and Hospital Authority (Other)
Collaborators: McNeil Consumer & Specialty Pharmaceuticals, a Division of McNeil-PPC, Inc. (Industry)
Responsible Party: Principal Investigator, Kennon Heard, Fellowship Director, Denver Health and Hospital Authority
Other Study IDs: COMIRB 09-0510
Record Dates: First submitted 2009-11-25; First posted 2009-11-30 (Estimated); Last update posted 2012-08-08 (Estimated); Status verified 2012-08

CONDITIONS: Acetaminophen-protein Adduct Formation
Keywords: acetaminophen; paracetamol; protein adduct; healthy volunteer; acetaminophen-protein adduct formation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Acetaminophen Group: Subjects who completed COMIRB 06-1265 and were assigned to the acetaminophen treatment group for that study.

SUMMARY:
The purpose of this study is to better understand the pharmacokinetics of acetaminophen and further clinical interpretations of laboratory results that confirm the presence of acetaminophen-cys adducts. This study will determine how long adducts persist in serum after a therapeutic course of acetaminophen as taken in a previous study (COMIRB 06-1265). Subjects will be asked to complete three study visits, each three days apart, following termination of COMIRB 06-1265. Each study visit will include collection of blood samples for batch testing of aminotransferase, serum acetaminophen and protein adducts. No interventions are planned.

ELIGIBILITY:
Inclusion Criteria:

* Any subject randomized to the acetaminophen arm of COMIRB 06-1265 and meets completion criteria

Exclusion Criteria:

* Subjects who enter the extended dosing period in protocol 06-1265.
* Subjects who were randomized to placebo.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All subjects who have met completion criteria for COMIRB 06-1265 and were assigned to the acetaminophen treatment group for that study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2009-11; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
The primary outcome of the proposed study is to determine the proportion of subjects with acetaminophen-cys adduct concentrations above the limit of quantification at day 6 after stopping maximum acetaminophen dosing. | Day 6

SECONDARY OUTCOMES:
The secondary outcomes of the proposed study are the serum acetaminophen-cys adduct concentrations at 3, 6, 9 days after stopping maximum acetaminophen dosing of the COMIRB 06-1265 study. | Days 3, 6, 9

CONTACTS AND LOCATIONS:
Overall Officials: Kennon Heard, MD, Principal Investigator — Denver Health and Hospital Authority
Locations (2):
- United States (2):
  - University of Colorado Hospital CTRC, Aurora, Colorado
  - Denver Health and Hospital Authority, Denver, Colorado